CLINICAL TRIAL: NCT00152009
Title: A Phase III, Randomized, Multi-Center, Double-Blind, Parallel-Group, Placebo-Controlled Safety and Efficacy Study of SPD503 in Children and Adolescents Aged 6-17 With Attention-Deficit/Hyperactivity Disorder (ADHD)
Brief Title: Safety and Efficacy of SPD503 in Treating Attention-Deficit/Hyperactivity Disorder (ADHD) in Children Aged 6-17
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPD503-301
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Results first posted 2009-11-26 (Estimated); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Attention Deficit Disorder With Hyperactivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Guanfacine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- SPD503 (Guanfacine HCl) (2 mg) (Experimental)
  Interventions: Drug: SPD503 (Guanfacine hydrochloride) (2 mg)
- SPD503 (3 mg) (Experimental)
  Interventions: Drug: SPD503 (3 mg)
- SPD503 (4 mg) (Experimental)
  Interventions: Drug: SPD503 (4 mg)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SPD503 (Guanfacine hydrochloride) (2 mg)
  Arms: SPD503 (Guanfacine HCl) (2 mg)
Drug: SPD503 (3 mg)
  Arms: SPD503 (3 mg)
Drug: SPD503 (4 mg)
  Arms: SPD503 (4 mg)
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and efficacy of SPD503 (Guanfacine hydrochloride) compared to placebo in the treatment of ADHD in children and adolescents aged 6-17

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a primary diagnosis of ADHD
* Male or non-pregnant female subject who agrees to comply with any applicable contraceptive requirements

Exclusion Criteria:

* Subject has current uncontrolled comorbid psychiatric diagnosis (except ODD) with significant symptoms
* History of seizure during the last 2 years
* Subject has any specific cardiac condition or family history of significant cardiac condition
* Subject is pregnant or lactating

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 345 (Actual)
Dates: Start 2003-01-29 (Actual); Primary Completion 2003-08-23 (Actual); Study Completion 2003-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda

REFERENCES:
- [Result] Biederman J, Melmed RD, Patel A, McBurnett K, Konow J, Lyne A, Scherer N; SPD503 Study Group. A randomized, double-blind, placebo-controlled study of guanfacine extended release in children and adolescents with attention-deficit/hyperactivity disorder. Pediatrics. 2008 Jan;121(1):e73-84. doi: 10.1542/peds.2006-3695. PMID 18166547
- See also: FDA recall information — http://www.fda.gov/opacom/7alerts.html
- See also: FDA-approved label — http://www.intuniv.com/documents/INTUNIV_Full_Prescribing_Information.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects were randomized to receive either 2, 3, or 4 mg SPD503 (Guanfacine hydrochloride) or placebo once-daily.
Groups:
- SPD503 2mg: Subjects were randomized to receive 2 mg SPD503 (Guanfacine hydrochloride) once-daily.
- SPD503 3mg: Subjects were randomized to receive 3 mg SPD503 (Guanfacine hydrochloride) once-daily.
- SPD503 4mg: Subjects were randomized to receive 4 mg SPD503 (Guanfacine hydrochloride) once-daily.
- Placebo: Subjects were randomized to receive Placebo once-daily.
Period: Overall Study
Arm/Group | SPD503 2mg | SPD503 3mg | SPD503 4mg | Placebo
Started | 87 | 86 | 86 | 86
Completed | 58 | 55 | 49 | 53
Not Completed | 29 | 31 | 37 | 33
Not completed — Adverse Event | 9 | 13 | 20 | 1
Not completed — Protocol Violation | 3 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 3 | 4 | 9
Not completed — Lost to Follow-up | 2 | 4 | 3 | 3
Not completed — Lack of Efficacy | 8 | 6 | 7 | 15
Not completed — ECG abnormalities | 2 | 2 | 2 | 1
Not completed — Sponsor's decision | 3 | 3 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SPD503 2mg | SPD503 3mg | SPD503 4mg | Placebo | Total
Number analyzed (Participants) | 87 | 86 | 86 | 86 | 345
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 87 | 86 | 86 | 86 | 345
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.6 (2.35) | 10.8 (2.76) | 10.1 (2.86) | 10.6 (2.70) | 10.5 (2.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 17 | 29 | 22 | 88
  Male | 67 | 69 | 57 | 64 | 257
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 87 | 86 | 86 | 86 | 345

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Attention Deficit Hyperactivity Disorder Rating Scale (ADHD-RS-IV) Score at Up to 5 Weeks
Description: Change in the Attention Deficit Hyperactivity Disorder Rating Scale-fourth edition (ADHD-RS-IV) total score from baseline. The ADHD-RS-IV consists of 18 items scored on a 4-point scale ranging from 0 (no symptoms) to 3 (severe symptoms) with total score ranging from 0 to 54.
Time Frame: Baseline and up to 5 weeks
Population: Intent to treat (ITT) defined as all subjects who were randomized to treatment and had the baseline and at least one post-randomization primary efficacy measurement.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | SPD503 2mg | SPD503 3mg | SPD503 4mg | Placebo
Number analyzed (Participants) | 84 | 82 | 81 | 78
Units on a Scale | -15.93 (1.37) | -16.03 (1.38) | -18.51 (1.39) | -8.51 (1.42)
Statistical Analysis 1: Comparison: SPD503 2mg vs Placebo; Test type: Superiority or Other; p = 0.0006, ANCOVA; Employed Dunnett's adjustment for multiple pairwise comparisons. Corresponding baseline efficacy scores obtained were used as covariates
Statistical Analysis 2: Comparison: SPD503 3mg vs Placebo; Test type: Superiority or Other; p = 0.0005, ANCOVA; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: SPD503 4mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]

2. Secondary Outcome: Change From Baseline in Conner's Parent Rating Scale-revised Short Version (CPRS-R) Score at Up to 5 Weeks
Description: The Conner's Parent rating Scale-revised short version (CPRS-R) consists of 27 questions graded on a scale from 0 (not true at all) reflecting no symptoms to 3 (very much true) reflecting severe symptoms with a total score ranging from 0 to 81. Higher scores are indicative of increased ADHD. This scale allows parents to respond on the basis of the child's behavior and help assess ADHD and evaluate problem behavior.
Time Frame: Baseline and up to 5 weeks
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | SPD503 2mg | SPD503 3mg | SPD503 4mg | Placebo
Number analyzed (Participants) | 66 | 61 | 58 | 65
Units on a Scale | -15.59 (1.86) | -15.43 (1.95) | -21.49 (2.00) | -8.66 (1.87)
Statistical Analysis 1: Comparison: SPD503 2mg vs Placebo; Test type: Superiority or Other; p = 0.025, ANCOVA; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: SPD503 3mg vs Placebo; Test type: Superiority or Other; p = 0.035, ANCOVA; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: SPD503 4mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Change From Baseline in Conner's Teacher Rating Scale-revised Short Version (CTRS-R) Score at Up to 5 Weeks
Description: The Conner's Teacher Rating Scale-revised short version (CTRS-R) consists of 28 questions graded on a scale from 0 (not true at all) reflecting no symptoms to 3 (very much true) reflecting severe symptoms with a total score ranging from 0 to 84. Higher scores are indicative of increased ADHD. This scale allows teachers to respond on the basis of the child's behavior and help assess ADHD and evaluate problem behavior.
Time Frame: Baseline and up to 5 weeks
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | SPD503 2mg | SPD503 3mg | SPD503 4mg | Placebo
Number analyzed (Participants) | 63 | 56 | 56 | 62
Units on a Scale | -13.02 (1.69) | -14.88 (1.79) | -15.26 (1.80) | -2.17 (1.70)
Statistical Analysis 1: Comparison: SPD503 2mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: SPD503 3mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: SPD503 4mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]

4. Secondary Outcome: Number of Participants With Improvement in Clinical Global Impression-Improvement (CGI-I)
Description: Clinical Global Impression-Improvement (CGI-I) consists of a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved) or 2 (much improved) on the scale.
Time Frame: up to 5 weeks
Population: ITT
Measure: Number; unit: Participants
Arm/Group | SPD503 2mg | SPD503 3mg | SPD503 4mg | Placebo
Number analyzed (Participants) | 84 | 82 | 81 | 78
Participants | 47 | 41 | 45 | 20
Statistical Analysis 1: Comparison: SPD503 2mg vs Placebo; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: SPD503 3mg vs Placebo; Test type: Superiority or Other; p = 0.0016, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: SPD503 4mg vs Placebo; Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel

5. Secondary Outcome: Number of Participants With Improvement in Parent Global Assessment (PGA)
Description: Parent Global Assessment (PGA) consists of a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved) or 2 (much improved) on the scale.
Time Frame: up to 5 weeks
Population: ITT
Measure: Number; unit: Participants
Arm/Group | SPD503 2mg | SPD503 3mg | SPD503 4mg | Placebo
Number analyzed (Participants) | 66 | 61 | 59 | 65
Participants | 41 | 31 | 39 | 15
Statistical Analysis 1: Comparison: SPD503 2mg vs Placebo; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: SPD503 3mg vs Placebo; Test type: Superiority or Other; p = 0.0013, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: SPD503 4mg vs Placebo; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel

6. Secondary Outcome: Change From Baseline in Child Health Questionnaire-Parent Form (CHQ-PF50) Score at 5 Weeks
Description: The Child Health Questionnaire-Parent Form (CHQ-PF50) was developed to measure the physical and psychosocial well-being of children aged 5 years of age and older. Total score ranges from 0-100. Increases in scores represent improved well-being in subjects as assessed by their parents.
Time Frame: Baseline and 5 weeks
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | SPD503 2mg | SPD503 3mg | SPD503 4mg | Placebo
Number analyzed (Participants) | 61 | 61 | 52 | 58
Units on a scale
  Psychosocial | 9.03 (1.22) | 9.01 (1.20) | 10.64 (1.32) | 5.72 (1.23)
  Physical | 0.24 (0.84) | -1.82 (0.84) | -2.13 (0.92) | -0.18 (0.86)
Statistical Analysis 1: Comparison: SPD503 2mg vs Placebo; Psychosocial category; Test type: Superiority or Other; p = 0.1438, ANCOVA; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: SPD503 3mg vs Placebo; Psychosocial category; Test type: Superiority or Other; p = 0.1426, ANCOVA; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: SPD503 4mg vs Placebo; Psychosocial category; Test type: Superiority or Other; p = 0.0191, ANCOVA; [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Arm/Group | SPD503 2mg | SPD503 3mg | SPD503 4mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/87 | 1/86 | 1/86 | 0/86
Other Adverse Events (participants affected / at risk) | 67/87 | 76/86 | 75/86 | 55/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SPD503 2mg (N=87) | SPD503 3mg (N=86) | SPD503 4mg (N=86) | Placebo (N=86)
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Asthma aggravated (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SPD503 2mg (N=87) | SPD503 3mg (N=86) | SPD503 4mg (N=86) | Placebo (N=86)
Abdominal pain upper (Gastrointestinal disorders) | 9 | 14 | 14 | 5
Dry mouth (Gastrointestinal disorders) | 2 | 8 | 5 | 1
Nausea (Gastrointestinal disorders) | 6 | 5 | 5 | 2
Fatigue (General disorders) | 16 | 18 | 13 | 3
Lethargy (General disorders) | 5 | 7 | 8 | 3
Pyrexia (General disorders) | 2 | 0 | 6 | 3
Upper respiratory tract infection (Infections and infestations) | 3 | 5 | 2 | 3
Appetite decreased (Metabolism and nutrition disorders) | 5 | 8 | 5 | 2
Dizziness (Nervous system disorders) | 4 | 5 | 9 | 2
Headache (Nervous system disorders) | 23 | 19 | 26 | 21
Sedation (Nervous system disorders) | 8 | 11 | 14 | 3
Somnolence (Nervous system disorders) | 21 | 29 | 33 | 3
Insomnia (Psychiatric disorders) | 5 | 7 | 5 | 4
Irritability (Psychiatric disorders) | 9 | 2 | 5 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 7 | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 5 | 3
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 3 | 5
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 5 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.